CLINICAL TRIAL: NCT05858190
Title: Comparison of Drug Eluting Balloon and Plain Old Balloon for the Treatment of Non-atherosclerotic Renal Artery Stenosis--A Protocol of a Multicenter Study
Brief Title: Drug-eluting Balloon for Treatment of Non-atherosclerotic Renal Artery Stenosis--a Multicenter Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS - 2133
Record Dates: First submitted 2023-04-05; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-03

CONDITIONS: Hypertension, Renovascular
MeSH Terms: conditions — Hypertension, Renovascular

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB group (Experimental): paclitaxel-coated balloon (Orchid, Acotec Scientific Holdings Limited, Beijing, China)
  Interventions: Procedure: Parallel Assignment
- POB group (Placebo Comparator)
  Interventions: Procedure: Parallel Assignment

INTERVENTIONS:
Procedure: Parallel Assignment — intervention group: treated with drug eluting balloon（paclitaxel-coated balloon； Orchid, Acotec Scientific Holdings Limited, Beijing, China)； control group :treated with plain old balloon

SUMMARY:
The study will test the efficacy of drug eluting balloon(DEB) for non-atherosclerotic renal artery stenosis. The DEB (paclitaxel eluting balloon) will be used in the intervention group, while the plain old balloon(POB) will be used in the control group. The primary outcome is the effect of blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

* age between 18y and 45y.
* with ≥ 60% stenosis in at least one renal artery.
* with hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg).
* patients with no severe renal insufficiency (eGFR>30 ml/min, length of the kidney ≥ 7cm).
* Good compliance.
* with informed consent.

Exclusion Criteria:

* With apparent atherosclerotic risk factors.
* With renal intervention or surgery history.
* With congenital anatomical anomaly.
* With severe renal insufficiency (length of the target kidney < 7cm, total
* eGFR<30ml/min, divided eGFR of the target kidney<8 ml/min)
* With contraindication for antiplatelet therapy.
* With severe cardiopulmonary insufficiency.
* Allergic to contrast medium
* Being pregnant or preparing for pregnancy
* With active cancer.
* Life expectancy < 12 month
* Without informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 9 months
  uninterrupted patency with no procedures performed on or at the margins of the treated segment or bypass

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song X, Fu Y, Lai Z, Di X, Zeng R, Shao J, Ni L, Liu Z, Song X, Ye W, Liu C, Liu B, Zheng Y, Chen Y. Drug-coated balloon for treatment of non-atherosclerotic renal artery stenosis-a multi-center study. BMC Cardiovasc Disord. 2023 Oct 16;23(1):510. doi: 10.1186/s12872-023-03484-5. PMID 37845604